CLINICAL TRIAL: NCT03640975
Title: Innate Lymphoid Cells in Eosinophilic Esophagitis (French Title : Cellules Lymphoïdes innées Dans l'Oesophagite à Eosinophiles)
Brief Title: Innate Immunity in Eosinophilic Esophagitis
Acronym: CLOE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17020JHLJ
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: eosinophilic esophagitis; children; innate immunity
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case : eosinophilic esophagitis: Children with symptoms suggestive of EoE and requiring an upper gastrointestinal endoscopy with biopsies of the esophageal mucosa
  Interventions: Other: Endoscopy
- control: Children in whom an endoscopy performed to explore symptoms of EoE revealed another condition (peptic oesophagitis, achalasia), or children in whom an endoscopy with biopsies has been performed to explore chronic abdominal or epigastric pain or suspected chronic inflammatory bowel disease
  Interventions: Other: Endoscopy

INTERVENTIONS:
Other: Endoscopy — The endoscopy will be performed under general anaesthesia using a flexible endoscope with an external diameter of between 4.9 and 9.2 mm, depending on the size of the child. In line with the guidelines, eight biopsies will be collected from the proximal, median and distal oesophagus for the routine analysis of esophageal remodelling and inflammation. Three of these biopsies will be used in the context of this study to analyse innate immune cells using flow cytometry and to determine the profile of cytokine expression. Two biopsies will be placed in sterile, 0.5 ml Nunc tubes containing a storage buffer (MACS® Tissue Storage Solution) and then stored in ice until the extraction of cells for cytometric analysis . The third specimen will be placed in a sterile tube and frozen immediately in liquid nitrogen for analyses of the esophageal microbiome.

SUMMARY:
The main aim of this study is to assess the expression of innate lymphoid cells in the esophageal mucosa of children with eosinophilic esophagitis (EoE) and in control subjects

DETAILED DESCRIPTION:
Children (aged 1 to 18 years) presenting with symptoms suggestive of EoE and requiring an upper gastrointestinal endoscopy with biopsies of the esophageal mucosa in order to confirm or exclude the diagnosis of EoE will be included.

Children paired for age in whom an endoscopy performed to explore symptoms of EoE revealed another condition (peptic oesophagitis, achalasia), or children paired for age in whom an endoscopy with biopsies has been performed to explore chronic abdominal or epigastric pain or suspected chronic inflammatory bowel disease, will be include as control subjects.

The endoscopy will be performed under general anaesthesia using a flexible endoscope with an external diameter of between 4.9 and 9.2 mm, depending on the size of the child. In line with the guidelines, eight biopsies will be collected from the proximal, median and distal oesophagus for the routine analysis of esophageal remodelling and inflammation. Three of these biopsies will be used in the context of this study to analyse innate immune cells using flow cytometry and to determine the profile of cytokine expression. Two biopsies will be placed in sterile, 0.5 ml Nunc tubes containing a storage buffer (MACS® Tissue Storage Solution) and then stored in ice until the extraction of cells for cytometric analysis. The third specimen will be placed in a sterile tube and frozen immediately in liquid nitrogen for analyses of the esophageal microbiome.

ILC1, 2 and 3 and their sub-types will be identified by means of structural criteria (size and granularity) and differential membrane and intracellular labelling using the specific markers shown below. All acquisitions and analyses will be achieved using a 13-colour NovoCyte cytometer (AACEA) and its associated software (NovoAxpressTM), which are available in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* children 1-18 years
* presenting with symptoms suggestive of EoE
* requiring an upper gastrointestinal endoscopy with biopsies of the esophageal mucosa in order to confirm or exclude the diagnosis
* Children paired for age in whom an endoscopy performed to explore symptoms of EoE revealed another condition (peptic oesophagitis, achalasia), or children paired for age in whom an endoscopy with biopsies has been performed to explore chronic abdominal or epigastric pain or suspected chronic inflammatory bowel disease, will be include as control subjects

Exclusion Criteria:

* immune deficiency
* auto immune diseases

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children presenting with symptoms suggestive of EoE and requiring an upper gastrointestinal endoscopy with biopsies of the esophageal mucosa
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
The numbers of innate immune cells | 1 year
  The counts of innate immune cells will be compared between EoE patients and controls

SECONDARY OUTCOMES:
Microbiota | 1 year
  Analyses of the composition of the esophageal microbiome will be performed using 16S rDNA sequencing after the extraction of DNA according to published protocols and/or using commercial kits (QlAamp DNA stool Mini Kit; QIAGEN). The pyrosequencing of 16S DNA, the identification of groups and phyla and initial biostatistical analyses will be carried out by specialised platforms.
Metabolomics | 1 year
  Metabolomic analyses will be performed on plasma and red blood cell extracts using a device such as an Orbitrap-Exactive equipped with an electrospray source. The data will be analysed using data processing tools available in the laboratory (software systems for signal detection and automatic alignment, annotation and statistical analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEZMI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker-Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No